CLINICAL TRIAL: NCT06769802
Title: The Effect of Using Nebula Bear on Anxiety and Fear During Nebulizer Application in Children: Randomized Controlled Trial
Brief Title: The Effect of Using Nebula Bear on Anxiety and Fear During Nebulizer Application in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Havva Nur Özlenir (Other)
Responsible Party: Sponsor-Investigator, Havva Nur Özlenir, Master Student/Nurse, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEUYLTEZ2024
Record Dates: First submitted 2024-12-31; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Children; Nebulizer Therapy
Keywords: Child; Nebulizer Therapy; Nebulizer; Nursing; Fear; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study was planned as a pre-test, post-test parallel group (invertion-control), randomized controlled experimental research type.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Nebula Bear Group (Experimental)
  Interventions: Behavioral: Experimental
- Active Comparator: Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Experimental — The children in this group and their mothers will be informed about the research and their written consent will be obtained. The scale will be filled in before the application. Before the application, Nebul will introduce the teddy bear to the mother and child. The teddy bear cannot be washed because it contains an electronic device. Therefore, it will be disinfected with a solution containing 60-70% alcohol before and after use. The recorded voice will then be played to the child and mother. Then, routine nebulizer treatment will be applied and the second audio recording will be played at the end of the treatment. The researcher will be with the child.
  At the end of the nebulizer treatment, after the mask is removed, the Child Fear Scale and the Child Anxiety Scale-State Scale will be filled out. The Child Fear Scale will be filled in by both the mother and the nurse and the average will be taken.
  Other Names: Nebula Bear Group
  Arms: Experimental: Nebula Bear Group
Behavioral: Control — The children in this group and their parents will be informed about the research and their written consent will be obtained. Scales will be filled in before application. Children in this group will receive routine nebulizer treatment and routine application will be performed. At the end of the treatment, the scales will be filled in again.
  Arms: Active Comparator: Control

SUMMARY:
Many respiratory system diseases are treated with inhalers. Providing inhaler treatment is provided by nebulizer devices. Taking the exact and effective dose of inhaler treatment affects the patient's recovery process. The use of nebulizer devices in children differs from that in adults. For children, the nebulizer may seem foreign and scary, which may cause them to reject inhaler treatment. Therefore, it is important to reduce anxiety and fear in children during nebulizer treatment. Since it is thought that the nebulizer bear, which is planned to be used in the study to reduce these negative situations caused by nebulizer treatment, may be effective in reducing anxiety and fear in children, it is thought that the study will have a positive physical and psychological contribution to children and parents.

DETAILED DESCRIPTION:
Especially in the first years of their lives, children are vulnerable to respiratory system diseases because their lungs and their relationships are adequately examined. The first 5 years of childhood are the period when the lower respiratory tract is at a high rate. It threatens all classified characteristics of lower respiratory tract diseases such as pneumonia and bronchiolitis, and is the most important cause of morbidity and mortality, especially for developmental diseases. Lower respiratory tract lines are recorded to be responsible for a large portion of emergency department visits and treatment admissions. Even in a developed country such as the United States, bronchiolitis occurs most commonly among young infants in a region. Pneumonia accounts for 13% of the cases seen in young children. The countries with the highest death rates were determined as the Central African Republic, Chad and Somalia. Moreover, with crowded populations and high mortality rates, it is known that almost one-third of lower respiratory tract infection deaths in children under 5 years of age occur in India and Nigeria. A systematic review of pneumonia in children noted aspects of serious illness in infants and young children and a high-range group, emphasizing that infants had a high initial recovery and hospitalization rate of pneumonia.It was reported that 13,800 children under the age of 5 died every day worldwide in 2020, and a total of 5 million children under the age of 5 died in the world in 2020. When the investigators look at the deaths caused by infectious diseases in Turkey, the investigators see that deaths caused by pneumonia and sepsis are at the forefront and the number of pneumonia cases doubled from 2016 to 2019.While respiratory tract infections are a major problem in children, the SARS-CoV-2 virus, which caused the Covid-19 infection that emerged in 2019 and affected the whole world, has caused high mortality rates in patients with severe disease, the elderly and patients with low immune systems. Administration of medication with nebulizers can be applied to all age categories, including children. Children's psychomotor skills vary depending on their developmental period and age. For this reason, there is no single type of nebula device that they can use in every period. When choosing a nebula device, the child's tolerance as well as his psychomotor skills should be taken into consideration. Effective treatment becomes difficult, especially in infants and children, due to the reactions observed during nebula intake. Multiple steps are required to use nebule devices correctly, and many children do not achieve adequate response to treatment because they cannot use the correct technique. Because children vary in their ability to cooperate with treatments, this can lead to significant dose changes and potentially affect the effectiveness of inhalation treatments. Being hospitalized and encountering unfamiliar equipment such as a nebulizer device can create fear and anxiety for the child. Children taking medication with a nebulizer can be aggressive, angry and resistant. Studies have found that 50% of babies and young children cry during inhaler therapy. Most pediatric procedures are traumatic, painful and stressful for children. Nurses should apply atraumatic care to minimize the traumatic effects of hospitalization on the child. In this context, it is important for pediatric nurses to reduce the child's stress, anxiety and fear during nebulizer application. The higher the child's anxiety, the less ability he or she will have to cope. Studies emphasize that it is important to encourage effective coping methods to minimize anxiety in children experiencing a medical condition.In a study by Zhang et al., where they investigated the effect of interactive play on children's aerosol therapy experience, compliance was found to increase significantly. Interactive games have been shown to clearly reduce tension in children and improve adherence to treatment. With the help of technology, games can be created to increase motivation and distract during treatment. A review of the literature shows that the age range of 6-12 is commonly considered and that the most used technologies are computer-based games and that games are generally designed to distract or motivate in physical rehabilitation. Robots, devices with hand-held interfaces and voice interactive technologies are still little used. In the study conducted by Logan et al. with an interactive SR teddy bear, it was found that children's joy and agreeableness levels were higher compared to a normal plush animal. A systematic review shows that the use of tangible interactive devices has decreased even more since 2011. However, recent research shows that toys with tangible user interfaces are more effective than traditional devices and even tactile handheld devices. Children are selective and eager to learn from others. When the studies on children's interaction with robots are examined; It shows that young children easily establish relationships with robots as guides in an unfamiliar environment. Combining physical spaces in a technological game is perceived as easier and more fun than screen-based activities. Concrete objects to be used in the game can be toys that children are familiar with. As a result, when the literature was examined, it was determined that nebulizer treatment caused anxiety and fear in children and it was seen that studies on this subject were needed. In the light of this information, a randomized controlled study was planned based on the studies in the literature. The aim of this study was to examine the effect of nebulizer treatment on anxiety and fear in children.

ELIGIBILITY:
Inclusion Criteria:

Are between the ages of 4-6, Parent's ability to read and write Turkish, Accompanied by their parents, Children who are willing to participate in the research will be included in the research, They receive the first nebule treatment of their hospitalization.

Exclusion Criteria:

Have mental disabilities or communication problems, Visual or hearing impairment, Those who have any body function deficiency Children who routinely use nebulizers

-

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Parent and Child Information Form | It will be filled out by the parent within the first 60 minutes of the child's hospitalization. (Approximately 5 minute.)
  Parent and child information form was created by researchers according to the literature. In the form content; It contains information about introductory characteristics about the child and the family (age, mother's education level, number of children, medical diagnosis, previous hospitalization, previous use of nebule therapy) and consists of 9 questions.
Child Fear Scale | It will be filled out by the researcher and parent 5 minutes before the procedure and 5 minutes after the procedure (Approximately 10 minute).
  This scale was used by McMurty et al.ild or the researcher to measure children's anxiety levels. It was developed by in 2011. The scale was developed by Gerçeker et al. in 2018. It has been validated in Turkish by and is aimed at children aged 4-10. Facial muscles changes in fearful expressions were drawn by a graphic designer based on photographs of frigtened faces. The scale can be used by the family, the child or the researcher to evaluate children. In this scale, the child is shown a scale containing five facial expressions rated between 0 and 4 points. While 0 indicates no fear and anxiety; 4 shows the highest fear and anxiety. These are: "0" neutral expression (no anxiety), "1" very little fear (very little anxiety), "2" some fear (some anxiety), "3" more fear (more anxiety), "4" the most fear possible. It is considered high fear (severe anxiety).
Children's Anxiety Meter-State (CAM-S) | It will be filled out by the child 5 minutes before the procedure and 5 minutes after the procedure (Approximately 5 minute).
  Children's Anxiety Meter-State was developed by Ersig et al. in 2013. A scale is a scale similar to a thermometer with horizontal lines. It is aimed at children aged 4-10 and was developed to measure children's anxiety. Teach kids: "Imagine all your anxious feelings are at the bottom." When instructed" If anxious feelings are high, paint the thermometer upwards with a pencil.Before filling out the scale, the child's number ordering level should be evaluated. Children who do not understand these instructions are not allowed to fill out the scale. After the child makes a rating on the scale, a transparent meter is placed on the scale and the marked point is measured.Half-point increments are rounded to the nearest number. The scale score is between 0-10.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No